CLINICAL TRIAL: NCT04549246
Title: Spatially Fractionated Radiation (Grid) Therapy for Tumors of the Head & Neck, Thorax, Abdomen, Pelvis, and Extremities
Brief Title: Grid Therapy for Tumors of the Head, Neck, Thorax, Abdomen, Pelvis and Extremities.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dawn M. Owen, M.D., Ph.D., Principal Investigator, Mayo Clinic
Other Study IDs: ROR1903; NCI-2022-105 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); ROR1903 (Other: Mayo Clinic Radiation Oncology); 19-012801 (Other: Mayo Clinic Institutional Review Board); 24-005944 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-08-13; First posted 2020-09-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Radiation Therapy Complication; Tumor Neck; Tumor Abdomen
MeSH Terms: conditions — Head and Neck Neoplasms; Abdominal Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Spatially Fractionated Radiation (GRID) Therapy — Grid therapy allows for high doses of radiation to be delivered over several spatially distinct, small regions. This permits regions of very high dose to a large tumor away from critical structures, which could be beneficial in both palliative and definitive treatments. Additionally, allowing for high doses to be delivered could pose a benefit for radioresistant histologies.

SUMMARY:
This study is an observational registry study evaluating the clinical outcomes of grid therapy. Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this study. Once consent has been obtained, baseline adverse event and QOL data will be collected and subjects will undergo grid therapy and follow-up at 2-4 weeks (for toxicity), and 3-6 months (for toxicities and radiographic control) then per clinical discretion up to 1 year. Patients will be evaluated according to the physician's standard practice and discretion. Patient data will be drawn from the patients' medical records and reported by means of a web-based electronic data collection (EDC) system. Patients will be considered "on study" until 60 months of observation has occurred, withdrawal of consent, lost to follow-up, or study closure. See below for the clinical visit flowchart for data collected at baseline and standard clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors of the head and neck, thorax, abdomen, pelvis, and extremities.
* Age ≥ 18 years.
* Histological confirmation of oncologic diagnosis.
* Completed oncologic imaging (per discretion of treating physician)
* ECOG Performance Status 0-3
* Ability to complete questionnaire(s) by themselves or with assistance.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Provide informed written consent.

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy. NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumors of the head, neck, thorax, abdomen, pelvis and extremities.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Local/radiographic control rate | 3-6 months
  Assessed according to Response Evaluation Criteria In Solid Tumors (RECIST), a standard system to measure how cancer responds to different treatments, including chemotherapy, immunotherapy, and radiation therapy. The local/radiographic control rate will be estimated overall and by palliative/definitive patient status in patients treated with grid therapy.

SECONDARY OUTCOMES:
To describe the adverse event profile (acute and late) of grid therapy by assessment of grade 3 or higher adverse events | through study completion, approximately 5 years
  Assessed by the number of grade 3 or higher adverse events (acute and late) that occur after grid therapy. Adverse events will be defined based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria.
Overall survival after grid therapy | through study completion, approximately 5 years
  Overall survival is defined as the length of time from either the date of diagnosis or the start of treatment that patients diagnosed with the disease are still alive.
Local/regional progression after grid therapy | through study completion, approximately 5 years
  Assessed by the number of patients to have local and/or regional progression after grid therapy. Local progression is defined as cancer recurring in the same place as the original cancer or very close to it. Regional progression is defined as cancer/tumor that has grown or spread into lymph nodes or tissues near the original cancer.
Recurrence rate | through study completion, approximately 5 years
  Number of patients to have tumor recurrence after grid therapy
Distant disease control | through study completion, approximately 5 years
  Distant disease control is defined as cancer that has spread from the original (primary) tumor to distant organs or distant lymph nodes.
Planning and delivery of grid therapy. | 5 years
  Total amount of time taken for planning and delivery of grid therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Owen, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials